CLINICAL TRIAL: NCT02188511
Title: Effects of Electronic Cigarettes on Lung Biology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 1312014623
Record Dates: First submitted 2014-07-02; First posted 2014-07-11 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Lung Disease; Lung Disorder
Keywords: E-Cigarettes; Lung; Non-Smokers; Lung Biology
MeSH Terms: conditions — Lung Diseases; Vaping | interventions — Electronic Nicotine Delivery Systems; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Experimental): Electronic cigarette (nicotine/placebo) - Day 8 Intervention: Electronic cigarette exposure will be limited to one day.
  Interventions: Other: Group A
- Group B (Experimental): Electronic cigarette (nicotine/placebo) - Days 7 through 8 Electronic cigarette exposure will be limited to two days
  Interventions: Other: Group B
- Group C (Experimental): Electronic cigarette (nicotine/placebo) - Days 6 through 8 Electronic cigarette exposure will be limited to 3 days
  Interventions: Other: Group C
- Group D (Experimental): Electronic cigarette (nicotine/placebo) - Days 5 through 8 Electronic cigarette exposure will be limited to 4 days
  Interventions: Other: Group D
- Group E (Experimental): Electronic cigarette (nicotine/placebo) - Days 4 through 8 Electronic cigarette exposure will be limited to 5 days.
  Interventions: Other: Group E

INTERVENTIONS:
Other: Group A — 90 minutes prior to the bronchoscopy on day 8, the subject will be asked to inhale 10 puffs of a Blu brand e-cigarette (for the nicotine-containing e-cigarette, this is approximately equivalent to < 1 cigarette). At 30 minutes prior to the bronchoscopy procedure if the subject has no adverse effect to the e-cigarette he/she will again be asked to inhale 10 puffs of the Blu e-cigarette.
  Other Names: Electronic cigarette (nicotine/placebo)- Day 8
  Arms: Group A
Other: Group B — On days 7 and 8, subjects will be asked to inhale 10 puffs of a Blu brand e-cigarette (90 minutes prior to bronchoscopy on day 8). If the subject has no adverse effect to the e-cigarette he/she will again be asked to inhale 10 puffs of the Blu e-cigarette an hour later (30 minutes prior to bronchoscopy on day 8).
  Other Names: Electronic cigarette (nicotine/placebo)- Days 7 and 8
  Arms: Group B
Other: Group C — On days 6 through 8, subjects will be asked to inhale 10 puffs of a Blu brand e-cigarette (90 minutes prior to bronchoscopy on day 8). If the subject has no adverse effect to the e-cigarette he/she will again be asked to inhale 10 puffs of the Blu e-cigarette an hour later (30 minutes prior to bronchoscopy on day 8).
  Other Names: Electronic cigarette (nicotine/placebo) - Days 6 through 8
  Arms: Group C
Other: Group D — On days 5 through 8, subjects will be asked to inhale 10 puffs of a Blu brand e-cigarette (90 minutes prior to bronchoscopy on day 8). If the subject has no adverse effect to the e-cigarette he/she will again be asked to inhale 10 puffs of the Blu e-cigarette an hour later (30 minutes prior to bronchoscopy on day 8).
  Other Names: Electronic cigarette (nicotine/placebo)- Days 5 through 8
  Arms: Group D
Other: Group E — On days 4 through 8, subjects will be asked to inhale 10 puffs of a Blu brand e-cigarette (90 minutes prior to bronchoscopy on day 8). If the subject has no adverse effect to the e-cigarette he/she will again be asked to inhale 10 puffs of the Blu e-cigarette an hour later (30 minutes prior to bronchoscopy on day 8).
  Exposure to e-cigarettes will be limited to the nicotine equivalent of 1/2 pack of cigarettes to mitigate the risk of addiction to nicotine.
  Other Names: Electronic cigarette (nicotine/placebo) - Days 4 through 8
  Arms: Group E

SUMMARY:
E-cigarettes are an increasingly popular alternate nicotine delivery system, but nothing is known about the effects of electronic cigarettes on the lungs. We hypothesize that e-cigarettes disorder airway epithelial and alveolar macrophages biology. Our goal is not to carry out a large epidemiologic study of electronic cigarette users to study lung function and other possible abnormal clinical phenotypes, but rather to focus on whether electronic cigarette smoke disorders the biology of the lung cells first exposed to the electronic cigarette smoke, a parameter that is the precursor of abnormalities in lung function and which is far more sensitive than lung function.

DETAILED DESCRIPTION:
The specific aim of this study is to assess the hypothesis that electronic smoking disorders the biology of the airway epithelium and alveolar macrophages, to evaluate these changes in the lungs of normal nonsmokers exposed to electronic cigarettes, and to directly determine if the inhaled smoke from electronic cigarettes disturbs the biology of the naïve lung that has not been exposed to tobacco products. Because nicotine can be addictive with continual use, we will limit the exposure to a maximum of a nicotine equivalent of 1/2 pack of cigarettes over a 5 day period, a level that has been used safely in studies of healthy nonsmokers' naïve to nicotine.

To obtain the most unbiased data about the effect of electronic cigarette use on the lung, normal nonsmokers will be briefly exposed to electronic cigarettes and lung cells, airway epithelium and alveolar macrophages, lung epithelial lining fluid (ELF) and serum will be collected before and after e-cigarette exposure. There will be 5 study groups consisting of 10 non-smoker subjects (A-E), with each group undergoing an increased exposure to the amount of e-cigarettes (Group a being the lowest exposure, group E being the highest). Six of the subjects in each group will be exposed to e-cigarettes with nicotine while the remaining four in each group being exposed to nicotine-free e-cigarettes. Subjects will be assigned to use electronic cigarettes that either do or do not contain nicotine in a randomized, blinded manner.

The duration of which the subjects will be observed for e-cigarette exposure will be 8 days. Baselines for each group will be established on Day 1 in which all subjects will undergo a bronchoscopy and an assessment of vital signs.

For subjects in group A, at the day 8 visit after the vital signs are assessed, 3 hours prior to bronchoscopy, the subject will be asked to inhale 10 puffs of a "Blu" brand e-cigarette (for the nicotine-containing e-cigarette, this is approximately equivalent to < 1 cigarette). At 2 hours prior to the bronchoscopy procedure, if the subject has no adverse effect to the e-cigarette he/she will again be asked to inhale 10 puffs of the "Blu" e-cigarette. The vital signs will again be confirmed and any symptoms assessed prior to proceeding with bronchoscopy. Subjects in group B will undergo an identical exposure, but on both days 7 and 8. Subjects in group C will undergo similar exposure on days 6-8, group D on days 5-8, and group E days 4-8 for a maximum of 5 exposure days prior to bronchoscopy. The research team will contact subjects at 1 month and 6 months after their Day 8 bronchoscopy in order to determine whether or not they have become dependent on nicotine.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 21 or older
* Must be capable of providing informed consent
* Self-reported never-smokers, with current smoking status validated by the absence of nicotine metabolites in urine (nicotine <2 ng/ml and cotinine <5 ng/ml)
* Normal physical examination
* Good overall health without history of chronic lung disease, including asthma, and without recurrent or recent (within 3 months) acute pulmonary disease
* Normal routine laboratory evaluation, including general hematologic studies, general serologic/immunologic studies, general biochemical analyses, and urine analysis
* Not taking any medications relevant to lung disease or having an effect on the airway epithelium
* Negative HIV serology
* Normal chest X-ray (PA and lateral)
* Normal electrocardiogram (sinus bradycardia, premature atrial contractions are permissible)
* Females - not pregnant
* No history of allergies to medications to be used in the bronchoscopy procedure
* Willingness to participate in the study

Exclusion Criteria:

* Unable to meet the inclusion criteria
* Current active infection or acute illness of any kind
* Evidence of malignancy within the past 5 years
* Current alcohol or drug abuse
* Pregnancy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Airway epithelium and aveolar macrophage | 8 days
  Changes in airway epithelium and aveolar macrophage will be measured by bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Staudt MR, Salit J, Kaner RJ, Hollmann C, Crystal RG. Altered lung biology of healthy never smokers following acute inhalation of E-cigarettes. Respir Res. 2018 May 14;19(1):78. doi: 10.1186/s12931-018-0778-z. PMID 29754582